CLINICAL TRIAL: NCT00998829
Title: An Australian Cross-Sectional Epidemiological Study To Evaluate The Prevalence Of Undiagnosed Psoriatic Arthritis In Psoriasis Patients In Dermatology Practice Focusing On Disease Severity, Disease Burden And Quality Of Life
Brief Title: Study Evaluating The Prevalence Of Undiagnosed Psoriatic Arthritis In Patients With Plaque Psoriasis
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0881A6-4611; B1801063
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: Arthritis, Psoriatic; Psoriasis
Keywords: psoriasis; psoriatic arthritis; epidemiology; prevalence
MeSH Terms: conditions — Arthritis, Psoriatic; Psoriasis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study population: The group comprises the entire study population
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — There is no therapeutic intervention in this study. However PASE (Psoriatic Arthritis Screening and Evaluation) and other patient questionnaires will be completed by participants.

SUMMARY:
This study aims to collect Australian data on the prevalence of undiagnosed psoriatic arthritis in patients with plaque psoriasis. In addition the study will assess disease severity and quality of life in Australian patients with psoriasis attending specialist dermatology clinics.

DETAILED DESCRIPTION:
Consecutive psoriasis patients seen at each site will be invited to participate in the study

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of plaque psoriasis
* >= 18 years of age
* Able to complete English-language questionnaires

Exclusion Criteria:

* Participation in an interventional clinical trial in previous 3 months
* Known rheumatologist-confirmed psoriatic arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Specialist dermatology clinics
Sampling Method: Probability Sample
Enrollment: 458 (Actual)
Dates: Start 2010-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the prevalence of undiagnosed psoriatic arthritis in patients presenting with plaque psoriasis using the PASE (Psoriatic Arthritis Screening and Evaluation) questionnaire based on a score of ≥ 44 on the questionnaire | 14 days
Evaluate the positive predictive value between PASE (Psoriatic Arthritis Screening and Evaluation) score ≥ 44 and rheumatologist-confirmed diagnosis of psoriatic arthritis in a population of tertiary Australian psoriasis patients | 14 days

SECONDARY OUTCOMES:
Evaluate the proportion of patients within the enrolled patient population with moderate-to-severe plaque psoriasis (PASI [Psoriasis Area and Severity Index] > 10) | 1 day
Evaluate the proportion of patients in a tertiary population with moderate-to-severe psoriasis with respect to treatment history and current treatment | 1 day
Describe quality of life (QoL) in a tertiary psoriasis patient population | 1 day
Explore the relationship between disease severity and QoL (quality of life) and stratified by the presence or absence of psoriatic arthritis in a tertiary population | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- Australia (9):
  - Pfizer Investigational Site, Camperdown, New South Wales
  - Pfizer Investigational Site, Darlinghurst, New South Wales
  - Pfizer Investigational Site, St Leonards, New South Wales
  - Pfizer Investigational Site, Westmead, New South Wales
  - Pfizer Investigational Site, Carina Heights, Queensland
  - Pfizer Investigational Site, Bedford Park, South Australia
  - Pfizer Investigational Site, Box Hill, Victoria
  - Pfizer Investigational Site, Fitzroy, Victoria
  - Pfizer Investigational Site, Parkville, Victoria

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0881A6-4611&StudyName=Study%20Evaluating%20The%20Prevalence%20Of%20Undiagnosed%20Psoriatic%20Arthritis%20In%20Patients%20With%20Plaque%20Psoriasis